CLINICAL TRIAL: NCT04842643
Title: A Phase 3, Open-label, Non-controlled, Multi-dose, Extension Study to Evaluate the Long-term Safety and Tolerability of IGSC, 20% in Japanese Subjects With Primary Immunodeficiency Disease (PID)
Brief Title: An Extension Study of TAK-664 for Japanese People With Primary Immunodeficiency Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-664-3002; U1111-1265-9447 (Other: WHO); jRCT2041210006 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-04-11; First posted 2021-04-13 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Primary Immunodeficiency Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGSC, 20% (Experimental): Participants who completed Epoch 2 of core study TAK-664-3001 (NCT04346108), received between 50 to 200 mg/kg of Immune globulin subcutaneous (IGSC) infusion, 20% infusion once a week (Epoch 2 regimen) and 100 to 400 mg/kg of IGSC infusion, 20% biweekly (Epoch 3 regimen) until the study drug becomes commercially available.
  Interventions: Biological: IGSC 20% infusion

INTERVENTIONS:
Biological: IGSC 20% infusion — IGSC 20% infusion,
  Other Names: Immune Globulin Infusion (Human)

SUMMARY:
This study is an extension study for participants with primary immunodeficiency disorders who were previously treated with IGSC, 20% in the TAK-664-3001 study. They must have completed that study or be about to complete it before joining this study. Participants will continue treatment with IGCS, 20% in this study.

The main aim of this study is to check for side effects from long-term treatment with IGSC, 20% . This medicine is not yet licensed in Japan, so participants will be treated with IGSC, 20% until it becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has completed or is about to complete Takeda Clinical Study TAK-664-3001.

   A participant is considered to have completed Study TAK-664-3001 successfully if they fulfill the following criterion: Completed Epoch 2, in which IGSC, 20% is administered weekly (completion of Epoch 3, in which IGSC, 20% is administered biweekly, is not mandatory for participation in TAK-664-3002 study).
2. Written informed consent is obtained from either the Participant or the Participant's legally authorized representative prior to any study-related procedures and study product administration.
3. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participant has developed a new serious medical condition during participation in Study TAK-664-3001 such that the Participant's safety or medical care would be impacted by participation in the extension study TAK-664-3002.
2. Participant is scheduled to participate in another non-Takeda clinical study involving an Investigational Product or device-used-in-clinical-trial in the course of this study.
3. If a female of childbearing potential, Participant is pregnant or has a negative pregnancy test but does not agree to employ adequate birth control measures for the duration of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Japan (8):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National defense medical college Hospital, Tokorozawa, Saitama
  - Kyushu University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Tokyo Medical Dental University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60769026688ad8001f42fb97

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Japan from 27 April 2021 to 25 April 2024.
Pre-assignment Details: Participants with primary immunodeficiency disorders who completed core study TAK-664-3001 (NCT04346108) were enrolled to receive Immune globulin subcutaneous (IGCS), 20 percent (%) in this current extension study (TAK-664-3002 [NCT04842643]). As per planned analysis, the data was collected, analyzed and reported for a single arm only and per dose level wise data was not collected in this study.
Groups:
- IGSC, 20%: Participants who completed Epoch 2 of core study TAK-664-3001 (NCT04346108), received between 50 to 200 mg/kg of IGSC infusion, 20% infusion once a week (Epoch 2 regimen) and 100 to 400 mg/kg of IGSC infusion, 20% biweekly (Epoch 3 regimen) until the study drug becomes commercially available.
Period: Overall Study
Arm/Group | IGSC, 20%
Started | 12
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All-Treated Set consisted of all enrolled participants who received IGSC, 20% administration at least once in this study.
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (21.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Non-serious TEAEs
Description: TEAEs were defined as adverse events (AEs) with onset after date-time of first dose of study drug (intravenous immunoglobulin [IGIV] or IGSC), or medical conditions present prior to the start of study drug (IGIV or IGSC) but increased in severity or relationship after date-time of first dose of study drug (IGIV or IGSC). A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Participants
  TEAEs | 12
  Serious TEAEs | 3
  Non-serious TEAEs | 12

2. Primary Outcome: Number of Participants With Drug-related and Non-related TEAEs
Description: TEAEs were defined as adverse events (AEs) with onset after date-time of first dose of study drug (intravenous immunoglobulin [IGIV] or IGSC), or medical conditions present prior to the start of study drug (IGIV or IGSC) but increased in severity or relationship after date-time of first dose of study drug (IGIV or IGSC). Any TEAE that was recorded by the investigator as "probably related" or "possibly related" to study drug was considered as study drug related AE, and any AE recorded as "unlikely related" or "not related" was considered as unrelated AE.
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Participants
  Drug-related TEAEs | 9
  Non-related TEAEs | 12

3. Primary Outcome: Number of Participants With Severe, Local and Systemic TEAEs
Description: A severe TEAE was an AE that caused considerable interference with the participant's usual activities. Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infusion site". Systemic TEAEs were defined as AEs that were not included in the Medical Dictionary for Regulatory Activities (MedDRA) Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site" or "infusion site".
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Participants
  Severe TEAEs | 3
  Local TEAEs | 8
  Systemic TEAEs | 12

4. Primary Outcome: Number of Participants With TEAEs Leading to Premature Discontinuation From Study and Infusion-associated TEAEs
Description: Infusion associated TEAEs were defined as any TEAE that began during study drug infusion or within 72 hours of completion of study drug infusion. TEAEs leading to premature discontinuation from study and infusion-associated TEAEs were reported.
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Participants
  TEAEs Leading to Premature Discontinuation | 0
  Infusion-associated TEAEs | 12

5. Secondary Outcome: Serum Trough Levels of Total Immune Globulin G (IgG) and IgG1, IgG2, IgG3, IgG4 Antibodies Subclasses Following Weekly Administration of IGSC, 20%
Description: Serum trough levels of total IgG and IgG1, IgG2, IgG3, IgG4 antibodies subclasses were determined by using standard assay methods.
Time Frame: At end of treatment in the current extension study TAK-664-3002 (i.e. 3 years)
Population: All-Treated Set consisted of all enrolled participants who received IGSC, 20% administration at least once in this study. Here" overall number of participants analyzed" signified participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: grams per liter (g/L)
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 5
grams per liter (g/L)
  IgG 1 | 6.14 [4.25 to 8.87]
  IgG 2 | 3.52 [2.35 to 5.28]
  IgG 3 | NA [NA to NA] — Geometric mean and 95% confidence interval (CI) could not be calculated because the values were below lower limit of quantification (LLOQ).
  IgG 4 | 0.305 [0.165 to 0.567]
  IgG Total | 11.0 [7.29 to 16.5]

6. Secondary Outcome: Serum Trough Levels of IgG and IgG1, IgG2, IgG3, IgG4 Antibodies Subclasses Following Biweekly Administration of IGSC, 20%
Description: Serum trough levels of IgG and IgG1, IgG2, IgG3, IgG4 antibodies subclasses were determined by using standard assay methods.
Time Frame: At end of treatment in the current extension study TAK-664-3002 (i.e. 3 years)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 7
g/L
  IgG 1 | 5.36 [4.55 to 6.33]
  IgG 2 | 3.42 [3.03 to 3.86]
  IgG 3 | NA [NA to NA] — Geometric mean and 95% CI could not be calculated because the values were below LLOQ.
  IgG 4 | 0.250 [0.219 to 0.284]
  IgG Total | 8.98 [7.78 to 10.4]

7. Secondary Outcome: Annual Rate of Validated Acute Serious Bacterial Infections (ASBI)
Description: The ASBI rate was calculated as the mean number of acute serious bacterial infections per participants per year. Annual rate of validated acute serious bacterial infections per participant was assessed. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: From first dose of study drug in core study TAK-664-3001 up to end of current extension study TAK-664-3002 (up to approximately 4.5 years)
Population: The Core Study All-Treated Set consisted of participants who received at least 1 dose of study drug (IGIV or IGSC) in TAK-664-3001.
Measure: Mean (Standard Deviation); unit: infections per year
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
infections per year | 0.00 (0.000)

8. Secondary Outcome: Annual Rate of All Infections
Description: The annual rate of infections was calculated as the mean number of infections per participant per year. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: infections per year
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
infections per year | 1.42 (1.119)

9. Secondary Outcome: Number of Days Participants Not Able to Attend School or Work to Perform Normal Daily Activities Due to Illness/Infection
Description: Number of days not able to attend school or work to perform normal daily activities due to illness/infection are standardized per year (365.25 days). Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
days | 1.91 [0.0 to 31.9]

10. Secondary Outcome: Number of Days Participants on Antibiotics
Description: Number of days on antibiotics was defined as the number of days those antibiotics were taken as concomitant medications and was standardized to per year (365.25 days). Number of days participants on antibiotics were reported. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
days | 2.55 [0.0 to 57.8]

11. Secondary Outcome: Number of Hospitalizations Due to Illness or Infection
Description: Number of hospitalizations were standardized to per year (365.25 days). Hospitalizations were measured by asking participants to report the number of nights they have stayed overnight in the hospital during the year, for something related to their own health. Number of hospitalizations due to illness or infection were reported. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hospitalization
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
hospitalization | 0.21 (0.370)

12. Secondary Outcome: Length of Hospital Stay Due to Illness or Infection
Description: Length of hospital stay per stay was standardized to per year (365.25 days). Number of days due to illness or infection were reported. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: The Core Study All-Treated Set consisted of participants who received at least 1 dose of study drug (IGIV or IGSC) in TAK-664-3001. Here" overall number of participants analyzed" signified participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 11
days | 0.00 [0.0 to 3.9]

13. Secondary Outcome: Number of Acute Physician Visits Due to Illness/Infection
Description: Number of acute physician visits is standardized to per year (365.25 days). Number of acute (urgent or unscheduled) physician visits due to illness/infection were reported. Reported timeframe included timeframe of core study TAK-664-3001 (NCT04346108) (Max approximately 1.5 year) and of current extension study (Max approximately 3 years) as data of this outcome measure was collected from first dose of core study to end of current extension study and the data is presented for participants who entered in current study from core study as per plan.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: visits per year
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
visits per year | 2.66 (2.652)

14. Secondary Outcome: Number of Participants With Their Response for Treatment Preference Questionnaire
Description: Treatment preference questionnaire is a self-administered questionnaire developed to assess participant's preference towards the administration of new IGSC therapy. There are 4-items on the questionnaire, which investigate a participant's preference on the clinic/hospital/home setting of receiving the immunoglobulin therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the IGSC treatment. For First question "Before participation in the trial(s), where did you receive your immunoglobulin therapy" participants were allowed to select multiple answers for options ("At the hospital"; "At home"; "Other") for their treatment. As a result, the sum of responders in the arm "IGSC, 20%: >=14 Years" for the first question were higher than the total number of participants analyzed in the category.
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: All-Treated Set consisted of all enrolled participants who received IGSC, 20% administration at least once in this study. As pre-specified in protocol, data was planned to be reported as per age criteria (2-13 years and >=14 years) for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- IGSC, 20%: 2-13 Years: Participants aged 2-13 years and who completed Epoch 2 of core study TAK-664-3001 (NCT04346108), received between 50 to 200 mg/kg of IGSC infusion, 20% infusion once a week (Epoch 2 regimen) and 100 to 400 mg/kg of IGSC infusion, 20% biweekly (Epoch 3 regimen) until the study drug becomes commercially available.
- IGSC, 20%: >=14 Years: Participants aged greater than or equal to (>=) 14 years and who completed Epoch 2 of core study TAK-664-3001 (NCT04346108), received between 50 to 200 mg/kg of IGSC infusion, 20% infusion once a week (Epoch 2 regimen) and 100 to 400 mg/kg of IGSC infusion, 20% biweekly (Epoch 3 regimen) until the study drug becomes commercially available.
Arm/Group | IGSC, 20%: 2-13 Years | IGSC, 20%: >=14 Years
Number analyzed (Participants) | 3 | 9
Participants
  Before participation in the trial(s), where did you receive your immunoglobulin therapy: At home | 0 | 0
  Before participation in trial(s), where did you receive your immunoglobulin therapy: At hospital | 3 | 8
  Before participation in the trial(s), where did you receive your immunoglobulin therapy: Other | 0 | 4
  Where do you Prefer to Receive Your Immunoglobulin Therapy: At Hospital | 1 | 1
  Where do you Prefer to Receive Your Immunoglobulin Therapy: At Home | 0 | 6
  Where do you Prefer to Receive Your Immunoglobulin Therapy: No Preference | 2 | 2
  The Frequency of Administration: Like very much | 1 | 1
  The Frequency of Administration: Like | 1 | 4
  The Frequency of Administration: No preference | 1 | 3
  The Frequency of Administration: Dislike | 0 | 1
  The Frequency of Administration: Dislike very much | 0 | 0
  The number of needlesticks per month: Like very much | 1 | 1
  The number of needlesticks per month: Like | 1 | 5
  The number of needlesticks per month: No preference | 1 | 2
  The number of needlesticks per month: Dislike | 0 | 1
  The number of needlesticks per month: Dislike very much | 0 | 0
  Total time spent for treatment per month: Like very much | 0 | 3
  Total time spent for treatment per month: Like | 1 | 2
  Total time spent for treatment per month: No preference | 1 | 1
  Total time spent for treatment per month: Dislike | 1 | 3
  Total time spent for treatment per month: Dislike very much | 0 | 0
  The ease of administration: Like very much | 1 | 3
  The ease of administration: Like | 2 | 4
  The ease of administration: No preference | 0 | 1
  The ease of administration: Dislike | 0 | 1
  The ease of administration: Dislike very much | 0 | 0
  The potential to self-administer: Like very much | 2 | 5
  The potential to self-administer: Like | 0 | 4
  The potential to self-administer: No preference | 0 | 0
  The potential to self-administer: Dislike: number analyzed (Participants) | 3 | 8
  The potential to self-administer: Dislike | 0 | 0
  The potential to self-administer: Dislike very much | 1 | 0
  Ability to fit treatment into schedule: Like very much | 1 | 5
  Ability to fit treatment into schedule: Like | 2 | 1
  Ability to fit treatment into schedule: No preference | 0 | 3
  Ability to fit treatment into schedule: Dislike | 0 | 0
  Ability to fit treatment into schedule: Dislike very much | 0 | 0
  The overall convenience: Like very much | 0 | 4
  The overall convenience: Like | 3 | 3
  The overall convenience: No preference | 0 | 2
  The overall convenience: Dislike | 0 | 0
  The overall convenience: Dislike very much | 0 | 0
  The amount of time administration takes: Like very much | 0 | 1
  The amount of time administration takes: Like | 1 | 5
  The amount of time administration takes: No preference | 1 | 1
  The amount of time administration takes: Dislike | 1 | 2
  The amount of time administration takes: Dislike very much | 0 | 0
  Complexity of administration: Like very much | 0 | 2
  Complexity of administration process: Like | 3 | 4
  Complexity of administration: No preference | 0 | 2
  Complexity of administration: Dislike | 0 | 1
  Complexity of administration: Dislike very much | 0 | 0
  Ability to self-administer: Like very much | 2 | 6
  Ability to self-administer: Like | 1 | 3
  Ability to self-administer: No preference | 0 | 0
  Ability to self-administer: Dislike very much | 0 | 0
  Ability to self-administer: Dislike | 0 | 0
  Choose to continue receiving IGSC: Yes | 3 | 7
  Choose to continue receiving IGSC: No | 0 | 2
  Factor influence decision: Two way needle, to see more variation in volume of chemical solution. | 0 | 1
  Factor influenced decision: Can be self-administered at home | 1 | 0
  Factor influenced decision: Easy administration method, easy to use | 0 | 1
  Factor influenced decision: Feel relieved | 0 | 1
  Factor influenced decision: Fewer side effects. IgG levels stabilized and became easier | 0 | 1
  Factor influence decision:.Take time to prepare, clean up, for area affected by needle to recover. | 0 | 1
  Factor influenced decision: Less susceptible to infections. Atopic dermatitis improved | 1 | 0
  Factor influenced decision: No answer | 1 | 0
  Factor influenced decision: No more coughing | 0 | 1
  Factor influenced decision: The values are stable | 0 | 1
  Factor influenced decision: Time is short | 0 | 1
  Factor influence decision: There were no major side effects and stable medical condition | 0 | 1

15. Secondary Outcome: Number of Participants With Tolerability Events Related to the Infusion of Study Drug
Description: An infusion was considered tolerable if the infusion rate was not reduced, or the infusion was not interrupted or stopped, due to a TEAE related to study drug infusion. A tolerability event was considered to have occurred if an infusion was not tolerable.
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Population: The Safety Analysis Set (SAS) consisted of all participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC, 20%
Number analyzed (Participants) | 12
Participants
  Infusion rate was reduced | 1
  Infusion was interrupted | 4
  Infusion was stopped | 1

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug in the current extension study TAK-664-3002, up to 3 years post-dose
Description: As per planned analysis, the data for this AE section was collected, analyzed and reported for a single arm only and per dose level wise data was not collected. All-Treated Set consisted of all enrolled participants who received IGSC, 20% administration at least once in this study.
Arm/Group | IGSC, 20%
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC, 20% (N=12)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC, 20% (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Administration site discolouration (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Asthenopia (Eye disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blepharitis (Eye disorders) | 2
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 5
Chills (General disorders) | 1
Chorioretinopathy (Eye disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Conjunctivitis (Infections and infestations) | 1
Conjunctivitis allergic (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cutaneous amyloidosis (Skin and subcutaneous tissue disorders) | 1
Cystitis (Infections and infestations) | 1
Dental caries (Gastrointestinal disorders) | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Gastroenteritis (Infections and infestations) | 3
Gingival pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 6
Heat illness (Injury, poisoning and procedural complications) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Influenza like illness (General disorders) | 1
Infusion site bruising (General disorders) | 1
Infusion site erythema (General disorders) | 1
Infusion site pain (General disorders) | 1
Infusion site pruritus (General disorders) | 1
Infusion site swelling (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site erythema (General disorders) | 3
Injection site haemorrhage (General disorders) | 1
Injection site pain (General disorders) | 3
Injection site reaction (General disorders) | 1
Injection site swelling (General disorders) | 4
Laryngitis (Infections and infestations) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Malaise (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Occult blood positive (Investigations) | 1
Oral herpes (Infections and infestations) | 2
Orthostatic intolerance (Nervous system disorders) | 1
Otitis externa (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Paronychia (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Pulpitis dental (Infections and infestations) | 2
Puncture site pain (General disorders) | 1
Pyrexia (General disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Retrograde amnesia (Nervous system disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rhinovirus infection (Infections and infestations) | 1
Seasonal allergy (Immune system disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2
Sinus headache (Nervous system disorders) | 1
Sinusitis (Infections and infestations) | 4
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Sudden hearing loss (Ear and labyrinth disorders) | 1
Tooth resorption (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vaccination complication (Injury, poisoning and procedural complications) | 5
Vaccination site joint erythema (General disorders) | 1
Vaccination site pain (General disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Wound (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT04842643/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04842643/SAP_001.pdf